CLINICAL TRIAL: NCT03126461
Title: Phase 2 Trial of SAbR Plus Ipilimumab Plus Nivolumab in Metastatic Melanoma Patients
Brief Title: SAbR Plus Ipilimumab Plus Nivolumab in Metastatic Melanoma Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the project was never initiated and no participants were enrolled, it was closed permanently
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU 082016-058
Record Dates: First submitted 2017-03-23; First posted 2017-04-24 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2018-04

CONDITIONS: Melanoma; Metastatic Melanoma
Keywords: metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SAbR plus ipilimumab plus nivolumab (Experimental): SAbR/GRID plus ipilimumab 3mg/kg IV q3wk x 4 plus nivolumab 1 mg/kg IV q3wk x 4, followed by nivolumab 240 mg IV q 2wk until progression or intolerable toxicity
  Interventions: Radiation: SAbR; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Radiation: SAbR — For patients treated on the "GRID A" regimen, a dose of 15-20 Gy will be delivered with the GRID device in either a single field, with prescription to dmax, or with parallel opposed GRID fields (matching beamlets from the opposed directions). For patients treated on the "GRID B" regimen, this same dose will be delivered, with a subsequent regimen of 3 Gy X 10 fractions, with the first of these fractions following the GRID dose.
  Other Names: Stereotactic ablative body radiation
Drug: Ipilimumab — ipilimumab 3mg/kg IV q3wk x 4
  Other Names: Yervoy®
Drug: Nivolumab — nivolumab 1 mg/kg IV q3wk x 4
  Other Names: Opdivo®

SUMMARY:
A one-arm, single center phase 2 trial of SAbR plus ipilimumab plus nivolumab in advanced metastatic melanoma patients

DETAILED DESCRIPTION:
SAbR/GRID plus ipilimumab 3mg/kg IV q3wk x 4 plus nivolumab 1 mg/kg IV q3wk x 4, followed by nivolumab 240 mg IV q 2wk until progression or intolerable toxicity

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of metastatic melanoma.
* Any number of prior systemic therapeutic regimens including chemotherapy, pathway inhibitors, biochemotherapy, investigational agents, and immunotherapies other than ipilimumab, nivolumab or other CTLA-4, PD-1 or PD-L1 inhibitors.
* Patients must have measurable disease in at least 2 non-radiated sites as defined by RECIST v1.1. All sites must be evaluated within 4 weeks prior to registration.
* Age ≥ 18 years.
* Eligible for SABR to 1-5 sites of disease (Refer to 3.2.10)
* Performance status ECOG 0-2.
* Adequate organ and marrow function as defined below:

  * leukocytes ≥ 1,000/mcL
  * absolute neutrophil count ≥ 1,000/mcL
  * platelets ≥ 75,000/mcl
  * total bilirubin < 2.5X institutional upper limit of normal or

    * 3 in subjects with Gilbert's Syndrome
  * AST(SGOT)/ALT(SPGT) ≤ 4 X institutional upper limit of normal
  * creatinine < 4X institutional upper limit of normal
  * hemoglobin >7g/dL
* Ability to understand and the willingness to sign a written informed consent.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of protocol treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* No concomitant therapy with any of the following: IL2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; or other investigational therapies; all such therapies must have been discontinued >4weeks prior to registration.
* No infection with HIV and no known history of hepatitis B or hepatitis C virus indicating acute or chronic infection or active TB.
* Patients are excluded if they have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated (Surgery or radiation) and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or localized adenocarcinoma of the cervix.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant or nursing.
* Patients are excluded if they have a history of prior treatment with ipilimumab, CTLA-4 inhibitor or agonist, nivolumab, PD-1 or PD-L1 inhibitor.
* Subjects who have had major surgery within 2 weeks prior to first dose of drug
* Subjects who have had radiation therapy within 2 weeks prior to first dose of drug
* Uncontrolled adrenal insufficiency or active chronic liver disease
* Any history of CNS metastases that is not adequately treated (surgery or radiation ) >14 days prior to registration.
* Any active known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose of study drug. Inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalent are permitted (although not encouraged) in the absence of active autoimmune disease.
* Subjects with life expectancy < 6 months
* Subjects receiving any other investigational or standard antineoplastic agents.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of tumor size from baseline to follow up | at 12, 24, 36 weeks
  treatment response rate-RR based on RECISTv1.1

SECONDARY OUTCOMES:
disease control rate | at 12, 24, 36 weeks
  disease control rate defined as response plus stable disease based on RECISTv1.1
Number of treatment-related adverse events | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
programmed death ligand-1 (PD-L1) expression | baseline, cycle 1 Day 1, and week 15
  compare tumor PD-L1 expression at 3 time points

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Albuquerque, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No